CLINICAL TRIAL: NCT01509131
Title: Low Volume Bowel Preparation for Colonoscopy: a Comparison Between PEG-CS Plus Bisacodyl Versus PEG-ASC
Brief Title: Evaluation of a Mixed Bowel Prep (2L PEG + Bisacodyl) Versus PEG With Ascorbate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promefarm S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMF105BC1/09
Record Dates: First submitted 2012-01-04; First posted 2012-01-12 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Bisacodyl; MoviPrep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2L PEG-CS plus bisacodyl (Experimental): Patients will be asked to take 2L PEG-CS plus bisacodyl (10-20 mg according to patient bowel habit)
  Interventions: Drug: 2L PEG-CS plus bisacodyl
- 2L PEG-ASC (Active Comparator): Patients will be asked to take PEG-ASC according to labeling instructions
  Interventions: Drug: 2L PEG-ASC

INTERVENTIONS:
Drug: 2L PEG-CS plus bisacodyl — Patients will be asked to take 2L of Lovolesse and bisacodyl (10-20 mg according to patient bowel habit)
  Other Names: Lovolesse 2L plus Lovoldyl 5 mg (2-4 tablets)
  Arms: 2L PEG-CS plus bisacodyl
Drug: 2L PEG-ASC — Patients will asked to take PEG-ASC according to labeling instructions
  Other Names: Moviprep
  Arms: 2L PEG-ASC

SUMMARY:
It is hypothesized that PEG 2L with citrate and simeticone plus bisacodyl will have similar bowel cleansing efficacy versus PEG 2L with ascorbate. Safety, tolerability, acceptance and compliance of the two reduced volume PEG-based bowel preparation will be also compared.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients undergoing a complete colonoscopy
* Patient written informed consent

Exclusion Criteria:

* Pregnant or lactating women or at a risk of becoming pregnant
* Hypersensitivity to any of the ingredients
* History of anaphylaxis to drugs or allergic reactions in general
* Known or suspected gastrointestinal obstruction or perforation
* Toxic megacolon; major colonic resection
* Heart failure (Class III or IV); severe renal failure; relevant diseases, that may interfere with the aim of the study
* Phenylketonuria;Glucose-6-phosphate dehydrogenase deficiency
* Unwillingness to co-operate and to comply with the requirements of the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quality of bowel preparation by BBPS | 20 minutes
  BBPS is an established rating scale to evaluate the quality of bowel preparation. A score greater than 6 is considered as success. The rate of success will be compared between the two groups.

SECONDARY OUTCOMES:
Difference in mucosal visibility between the two groups | 20 minutes
  Three point rating scale(0-2).
Number of patients with adverse events | 24 hours
  Patient questioning.
Difference in tolerability between the two groups | 24 hours
  Difference in the percentage of patients in the two groups who developed GI symptoms related to bowel preparation.
Difference in patients acceptability between the two groups | 24 hours
  Difference in the percentage of patients in the two groups who were willing to repeat the preparation and easy to take the bowel preparation.
Difference in patients compliance between the two groups | 24 hours
  Difference in the percentage of patients who took at least 75% of bowel preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — IRCSS Istituto Clinico Humanitas, Rozzano (MI) - Italy; Renzo Cestari, Prof. MD, Principal Investigator — Spedali Civili di Brescia, Brescia - Italy; Cesare Hassan, MD, Principal Investigator — Nuovo Regina Margherita, Roma - Italy; Angelo Andriulli, MD, Principal Investigator — IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo - Italy; Vito Annese, MD, Principal Investigator — Ospedale Careggi, Firenze - Italy
Locations (5):
- Italy (5):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - IRCCS Humanitas, Rozzano, Milano
  - Spedali Civili, Brescia
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Nuovo Regina Margherita, Roma